CLINICAL TRIAL: NCT02640014
Title: Specific Oral Immunotherapy in Food Allergy - Real-life Long-term Follow up (After Milk Oral Immunotherapy), Effect on Health-related Quality of Life and Cost-utility Analyses
Brief Title: Oral Immunotherapy in Food Allergy in Finland
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Tiina Kauppila, MD, MD, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1020AL001
Record Dates: First submitted 2015-12-17; First posted 2015-12-28 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Food Hypersensitivity; Immune System Diseases; Anaphylaxis
Keywords: Food allergy; Health-related quality of life (HRQL); Quality-adjusted life-years (QALYs); Oral immunotherapy (OIT); Cow´s milk allergy (CMA); Milk oral immunotherapy (MOIT)
MeSH Terms: conditions — Food Hypersensitivity; Immune System Diseases; Anaphylaxis | interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study 1: Milk OIT follow up (Experimental): Follow up on patient with severe milk allergy how have participated to milk OIT.
  Interventions: Dietary Supplement: Milk
- Study 1: Follow up (No Intervention): Follow up on patient with severe milk allergy how have not participated to milk OIT.

INTERVENTIONS:
Dietary Supplement: Milk — Milk Oral immunotherapy
  Arms: Study 1: Milk OIT follow up

SUMMARY:
The outcomes of oral immunotherapy (OIT) in food allergy study will provide more knowledge of oral immunotherapy. So far the OIT has showed in clinical experiments to be a interesting way to increase the unresponsiveness in severe food allergies. However little is known about it´s long-term outcomes, immunological mechanisms and there are no previous studies about cost-utility of OIT.

DETAILED DESCRIPTION:
The purpose of the present study is to examine the outcomes of the food oral immunotherapy on patients with severe food allergy in the three different subprojects:

Study 1: Long-term follow up after milk oral immunotherapy. The measured outcomes are long-term effectiveness (e.g. health-related quality of life), safety of desensitization and immunological changes.

Study 2: Measure health-related quality of life with disease-specific and generic questionnaire. The aim of this study is to define the suitability of the FAQLQ and the 15-D questionnaires for the Finnish food allergic patients. Another purpose of this study is to examine the relationship between FAQLQ and 15-D questionnaires.

Study 3: QALYs. This is called the cost-utility analyses and QALYs and its purpose is to calculate the cost of OIT and to define the cost-effectiveness of OIT by measuring QALYs. To our knowledge this will be the first pilot study to define the QALYs in food oral immunotherapy. The aim is to have 50-100 patients. The literature in other areas of medicine 50-100 patients in QALY-publishing is quite plain.

ELIGIBILITY:
Inclusion Criteria:

* Study 1: All the children have been eligible to participate milk OIT during the years 2005-2015.
* Study 2 + 3: Patients will start OIT treatment (to milk / egg / peanut).

Exclusion Criteria:

* Not willing to participate
* Active asthma, low lung function, pregnancy, cardiovascular or other disease that might worsen during the OIT.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-12; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Long-term effectiveness as a measure of milk consumption (dl/day). | Ten years
  Consumption of milk (dl/day)

SECONDARY OUTCOMES:
General health-related quality of life | One year
  To measure health-related quality of life by using a generic (Finnish 15-D questionnaire) before and one year after OIT.
Disease specific health-related quality of life | One year
  To measure health-related quality of life by using a disease specific questionnaires (Food Allergy Quality of Life Questionnaires, FAQLQ) before and one year after OIT.
Cost-utility analysis and health benefits by measuring quality-adjusted life-years (QALYs). | One year
  A Pilot study to define the cost of OIT and define the cost of quality-adjusted life-years (QALYs) with generic health-realted quality of life scale 15-D-questionnaire.
Incidence of Treatment - Emergent Adverse Events | Ten years
  Severe adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mika J Mäkelä, MD, PhD, Study Director — Chief Physician, Helsinki University Hospital
Locations (1):
- Helsinki University Central Hospital, Skin and Allergy Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kauppila TK, Hinkkanen V, Savinko T, Karisola P, Kukkonen AK, Paassilta M, Pelkonen AS, Makela MJ. Long-term changes in milk component immunoglobulins reflect milk oral immunotherapy outcomes in Finnish children. Allergy. 2023 Feb;78(2):454-463. doi: 10.1111/all.15479. Epub 2022 Aug 20. PMID 35969113